CLINICAL TRIAL: NCT06380647
Title: Comparison of Prophylactic Acyclovir and Placebo in Prevention of Eczema Herpeticum in Pediatric Burns
Acronym: childburn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Sharif, PROFESSOR, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0004
Record Dates: First submitted 2024-03-31; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Herpes Virus Infection
Keywords: Eczema herpeticum; pediatric burns; Acyclovir; Prophylaxis
MeSH Terms: conditions — Herpesviridae Infections; Kaposi Varicelliform Eruption

STUDY DESIGN:
Intervention Model Description: Sample size of 64 patients (32 patients in each group) was estimated by using 5% level of significance, 90% power of test with expected percentage of patients given prophylactic acyclovir as 81.3% and patients given placebo as 42.9%.
Who Masked: Participant
Masking Description: parents were blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A(32 patients) (Experimental): Group A patients were given intra venous acyclovir at dosage of 5-10 mg/kg/day into three doses for 7-14 days during their stay.Giant smear testing was done from suspected lesion on burn area to confirm viral infection
  Interventions: Drug: Intravenous Acyclovir
- Group B (32 patients) (Placebo Comparator): Group B patients were given intravenous normal saline 5-10 mg/kg into three doses as placebo for 7 to 14 days,Giant smear testing was done from suspected lesion on burn area to confirm viral infection
  Interventions: Drug: Intravenous Acyclovir

INTERVENTIONS:
Drug: Intravenous Acyclovir — Patients were observed for developing signs of eczema herpeticum and Tzanck smear was done every 10th day and first follow up at OPD after 7days of discharge following ward management protocol. If prophylactic acyclovir was efficacious then no eczema herpeticum developed. Patients who develop eczema herpeticum were isolated and were treated with injection acyclovir 15 to 30 mg/kg/day into three divided doses for 10 to 14 days.

SUMMARY:
Introduction: Early detection is important in treating patients with Eczema Herpeticum (EH), which may arise in paediatric burn patients. As soon as a clinical diagnosis is confirmed, antiviral medications should be started to ensure an early resolution of the disease. Several studies have indicated that acyclovir is the best treatment for EH lesions in the majority of individuals.

Objective: Compare efficacy of the prophylactic acyclovir and placebo in preventing eczema Herpeticum in paediatric burn patients

DETAILED DESCRIPTION:
Materials and Methods Study design: Randomised control trial. Setting: Pediatric burn unit Mayo hospital Lahore Duration: 1st October 2019 to 30th September 2020. Data collection procedure: All the patients were managed with intravenous fluids, antibiotics, antipyretics and hydrocolloid dressing as per ward routine management protocol along with prophylactic acyclovir and placebo. On the zero day of admission, after parents provided informed consent, patients were randomly assigned to one of two groups using a computer-generated table. Group A patients were given intra venous acyclovir divided into three doses for 7 to 14 days during their stay. Group B patients were given 15% intravenous Hypertonic sodium chloride divided into three doses as placebo for 7 to 14 days, so that parents could be blinded to group allocation. Patients were observed for developing signs of eczema Herpeticum and Tzanck smear was done every 10th day and first follow up at outpatient department after 7days of discharge.

ELIGIBILITY:
* age 1 month to ≤ 13 years .10 to 60 percent total body surface area (TBSA) burn.
* 2nd and 3rd degree burn Exclusion Criteria

  * Patients having previous history of skin disease.
  * Patients having any Comorbidity e.g. Psoriasis, asthma, atopic dermatitis and conjunctivitis.
  * Immunocompromised patients.
  * Patients on steroids or chemotherapy.
  * Patients already having eczema Herpeticum and positive baseline Tzanck smear

Ages: 1 Month to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with positive Tzanck smear | 1 year
  Prophylactic acyclovir was compared with placebo regarding preventing eczema herpeticum prophylactically

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sharif, Study Chair — King edward Medical University/Mayo Hospital Lahore
Locations (1):
- department of pediatric surgery King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
will be shared on request